CLINICAL TRIAL: NCT02741193
Title: Validation of Presurgical Motor Mapping With Transcranial Magnetic Stimulation (TMS) in Patients With Epilepsy
Brief Title: Presurgical Motor Mapping With Transcranial Magnetic Stimulation (TMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-00176
Record Dates: First submitted 2016-04-08; First posted 2016-04-18 (Estimated); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
Keywords: Transcranial magnet stimulation (nTMS); Brainsight Neuronavigation; Electromyography; EMG
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- nTMS (Experimental): Patients will receive a single-pulse TMS mapping of the motor area for the following reasons to determine the motor threshold, measure concurrent EMG, and mapping of the upper extremity.
  Interventions: Device: The Magstim Rapid2,

INTERVENTIONS:
Device: The Magstim Rapid2, — Transcranial Magnetic Stimulation, which is a microprocessor-controlled machine which delivers both single and repetitive transcranial magnetic stimulation (TMS).
  single and repetitive transcranial magnetic stimulation (TMS). TMS will be applied as single pulses to determine motor evoked potentials (MEPs), there will be no modulation of cortical excitability.

SUMMARY:
The aim of the study is to examine the degree of concordance between presurgical neuronavigation guided TMS (nTMS) and direct cortical stimulation (DCS) in identifying hand motor cortex in adults undergoing epilepsy surgery.

Navigated transcranial magnet stimulation (nTMS), MagStim RapidStim2 Magnetic stimulation will be delivered to hand primary motor cortex, with positive and negative functional sites determined through surface electromyography (EMG).

The study will involve patients ages 12-60 years, with planned neurosurgery involving implantation of intracranial subdural electrodes including over the precentral gyrus.

Navigated transcranial magnet stimulation (nTMS), MagStim RapidStim2 Magnetic stimulation will be delivered to hand primary motor cortex, with positive and negative functional sites determined through surface electromyography (EMG).

The primary outcome measure will be spatial correlation between topographic maps of hand motor representation obtained through nTMS compared to direct, extra-operative cortical stimulation performed as part of routine clinical care. A secondary outcome measure will be safety and tolerability of TMS in the epilepsy patients.

DETAILED DESCRIPTION:
This study will be an open-label feasibility study which applies nTMS to subjects with incoming epilepsy surgery and pre-surgical motor mapping. No study-related medication changes are expected -- participants will remain compliant with their regular anticonvulsant regimen throughout each study phase. All patients will have undergone a complete history and neurological exam as part of their routine clinical care at the New York University (NYU) Comprehensive Epilepsy Center.

Fourteen (14) patients will undergo epilepsy surgery with expected subdural grid coverage over primary motor cortex. Potential subjects will be identified at the weekly multi-disciplinary epilepsy conference. Subjects must have a recent (<2 years) MRI scan, and registration of the TMS coil to the MRI scan via the Brainsight neuronavigation system will be utilized to guide TMS coil placement (Gugino et al 2001). When a presurgical fMRI (functional magnetic resonance imaging) is available which demonstrates the patient's hand knob, the fMRI will be used with the Brainsight neuronavigation system. Subjects will be recruited and consented during a presurgical clinical visit where the patient's primary epileptologist will introduce members of the research team.

nTMS mapping

Patients will receive a session of single-pulse TMS mapping of the motor area, at the outpatient TMS clinic at NYU Neurology Ambulatory Care Center, at 240 E 38th St 20th Floor prior their epilepsy surgery according to the following procedures:

1. Determination of the motor threshold by (1) finding the most excitable region in the hand knob which elicits the strongest compound muscle action potential (CMAP) in the APB muscle; (2) finding the motor threshold by determining output stimulation intensity which generates peak to peak CMAP response above 50 mV (Millivolts) in 5/10 stimulation cycles (Rossini et al., 1994).
2. Concurrent EMG will be measured with electrodes placed at APB (abductor policis brevis atrial premature beat), abductor digiti minimi, flexor carpiradialis muscles. Reference electrode will be placed at the ipsilateral elbow above the brachial biceps muscle.
3. Mapping of the upper extremity. After determination of the MT (motor threshold), mapping of the UE(Upper Extremity) will be performed at 110% of the rMT (resting motor threshold). All positive and negative stimulation sites will be recorded and saved. Patients will be closely monitored during TMS stimulation. Each subject will have a complete neurological examined by a neurologist before and immediately after nTMS. Patients will also be provided a side effects questionnaire after TMS mapping. Patients will then be asked to keep a 7 day seizure diary after the nTMS session.

After epilepsy surgery patients will receive the standard care for post-operative patients which including close monitoring in ICU overnight. Patients will be transferred to the floor for further clinical evaluation before discharge. Clinical outcome will be evaluated in the post-operative clinic visit within 1 month after discharge. The value of a clinical follow up is to evaluate for any discrepancy between nTMS and DCS, to determine which modality better predicts functional outcome. Any seizure recurrence or neurological deficit will be recorded at the follow-up clinical visit.

The trial is designed to detect strength of spatial correlation between topographic maps of hand motor representation obtained through noninvasive nTMS compared to direct, extra-operative cortical stimulation obtained as part of usual clinical evaluation during epilepsy surgery, as measured by (a) average distance between positive motor mapping sites of DCS compared to nTMS and (b) degree of concordance between positive and negative motor mapping sites between DCS and nTMS, to generate positive and negative predictive values, and (c) average distance between positive motor functional sites of fMRI compared to nTMS.

ELIGIBILITY:
Inclusion Criteria:

* 12-60 years of age
* Planned neurosurgery involving implantation subdural electrodes over the precentral gyrus

Exclusion Criteria:

* Inability to sign informed consent .
* Hemiparesis worse than 4-/5 on the side contra lateral to the planned implant
* Inability to get an MRI, or MRI older than 2 years
* Frequent (>1 per day) motor seizures
* Prior neurosurgery
* Metal in the head, including shrapnel
* Implanted stimulation devices, including DBS (Deep Brain Stimulator), RNS (Responsive Neurostimulator), VNS (Vagus Nerve Stimulator), PPM (Permanent Pacemaker)
* Pregnancy
* Use of a medication known to increase the risk of seizures, including certain antipsychotics (clozapine), bronchodilators (aminophylline, theophylline), immunomodulatory agents (cyclosporine), and antibiotics (penicillins, cephalosporins, amphotericin, imipenem)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, MA, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- nTMS: Patients will receive a single-pulse TMS mapping of the motor area for the following reasons to determine the motor threshold, measure concurrent EMG, and mapping of the upper extremity.
  The Magstim Rapid2,: Transcranial Magnetic Stimulation, which is a microprocessor-controlled machine which delivers both single and repetitive transcranial magnetic stimulation (TMS).
  single and repetitive transcranial magnetic stimulation (TMS). TMS will be applied as single pulses to determine motor evoked potentials (MEPs), there will be no modulation of cortical excitability.
Period: Overall Study
Arm/Group | nTMS
Started | 2
Completed | 0
Not Completed | 2
Not completed — Participant deemed not to be a surgical resection candidate | 1
Not completed — Participant found to be seizure-free due to new epilepsy medication, did not participate | 1

BASELINE CHARACTERISTICS:
Population: No participants completed the trial nor had baseline characteristic data recorded.
Arm/Group | nTMS
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Average Distance Between Positive Motor Mapping Sites of DCS
Time Frame: 30 minutes
Population: No participants had data collected for this outcome measure.
Arm/Group | nTMS
Number analyzed (Participants) | 0

2. Primary Outcome: Average Distance Between Positive Motor Mapping Sites of nTMS
Time Frame: 30 minutes
Population: No participants had data collected for this outcome measure.
Arm/Group | nTMS
Number analyzed (Participants) | 0

3. Primary Outcome: Average Distance Between Positive Motor Functional Sites of fMRI
Time Frame: 30 minutes
Population: No participants had data collected for this outcome measure.
Arm/Group | nTMS
Number analyzed (Participants) | 0

4. Primary Outcome: Average Distance Between Positive Motor Functional Sites of nTMS
Time Frame: 30 minutes
Population: No participants had data collected for this outcome measure.
Arm/Group | nTMS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 minutes.
Arm/Group | nTMS
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02741193/Prot_SAP_000.pdf